CLINICAL TRIAL: NCT04921371
Title: Six Week Safety and Clinical Efficacy of Experimental Mouth Rinses: Effect on Gingivitis and Plaque
Brief Title: Six Week Study of Experimental Mouth Rinses: Effect on Gingivitis and Plaque
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCSORC001793; CCSORC001793 (Other: Johnson & Johnson Consumer Inc.)
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Gingivitis; Plaque
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy Reference Group (Other): Participants who are identified as healthy will be a comparison group. This group will participate in the examinations and plaque sampling only and will not receive a prophylaxis or product.
  Interventions: Other: Colgate® Cavity Protection Toothpaste; Other: Concept Curve Winter Series Toothbrush
- 5% Hydroalcohol Mouthrinse (Negative control) (Experimental): Participants after brushing with Colgate® Cavity protection toothpaste and Concept Curve winter series toothbrush will rinse mouth for 30 seconds with 20 milliliter (mL) of 5 percent (%) Hydroalcohol Mouthrinse twice daily (morning and evening) up to 6 weeks.
  Interventions: Other: Colgate® Cavity Protection Toothpaste; Other: Concept Curve Winter Series Toothbrush; Other: 5% Hydroalcohol Mouthrinse
- Listerine® Cool Mint® (Positive control) (Experimental): Participants after brushing with Colgate® Cavity protection toothpaste and Concept curve winter series Toothbrush will rinse mouth for 30 seconds with 20 mL of Listerine® Cool Mint® twice daily (morning and evening) up to 6 weeks.
  Interventions: Other: Colgate® Cavity Protection Toothpaste; Other: Listerine® Cool Mint®; Other: Concept Curve Winter Series Toothbrush
- Mouthrinse Prototype 1 (Experimental): Participants after brushing with Colgate® Cavity protection toothpaste and Concept Curve winter series toothbrush will rinse mouth for 30 seconds with 20 mL of Mouthrinse Prototype 1 twice daily (morning and evening) up to 6 weeks.
  Interventions: Other: Colgate® Cavity Protection Toothpaste; Other: Concept Curve Winter Series Toothbrush; Other: Mouthrinse Prototype 1
- Mouthrinse Prototype 2 (Experimental): Participants after brushing with Colgate® Cavity protection toothpaste and Concept Curve winter series toothbrush will rinse mouth for 30 seconds with 20 mL of Mouthrinse Prototype 2 twice daily (morning and evening) up to 6 weeks.
  Interventions: Other: Colgate® Cavity Protection Toothpaste; Other: Concept Curve Winter Series Toothbrush; Other: Mouthrinse Prototype 2

INTERVENTIONS:
Other: Colgate® Cavity Protection Toothpaste — Participants will use Colgate® Cavity protection toothpaste for brushing teeth twice daily.
Other: Listerine® Cool Mint® — Participants will use 20 mL of Listerine® Cool Mint® mouth rinse for 30 seconds after brushing twice daily.
  Arms: Listerine® Cool Mint® (Positive control)
Other: Concept Curve Winter Series Toothbrush — Participants will brush twice daily for 1 minute with the toothpaste and soft bristled toothbrush provided.
Other: 5% Hydroalcohol Mouthrinse — Participants will use 20 mL of 5% Hydroalcohol Mouthrinse for 30 seconds after brushing twice daily.
  Arms: 5% Hydroalcohol Mouthrinse (Negative control)
Other: Mouthrinse Prototype 1 — Participants will use 20 mL of Mouthrinse Prototype 1 for 30 seconds after brushing twice daily.
  Arms: Mouthrinse Prototype 1
Other: Mouthrinse Prototype 2 — Participants will use 20 mL of Mouthrinse Prototype 2 for 30 seconds after brushing twice daily.
  Arms: Mouthrinse Prototype 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of experimental mouth rinse formulations compared to a positive control mouth rinse and a hydroalcohol control mouth rinse for the reduction of gingivitis and plaque when used as an adjunct to tooth brushing during a six-week product usage period.

ELIGIBILITY:
Inclusion Criteria:

* Adequate oral hygiene (That is brush teeth daily and exhibit no signs or oral neglect)
* A minimum of 20 gradable teeth including 4 molars with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, teeth with veneers, or third molars will not be included in the tooth count
* A mean gingival index greater than or equal to (>=) 1.95 per the Modified Gingival Index at Baseline (for those in the randomized treatment group)
* A mean gingival index less than or equals to (<=) 0.75 per the Modified Gingival Index at Baseline (for those in the healthy reference group)
* A mean plaque index >= 1.95 per the 6 site Turesky modification of the Quigley-Hein Plaque Index at Baseline (for those in randomized treatment groups)
* Greater than or equal to 10 percent (%) bleeding sites at baseline (for those in randomized treatment groups)

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouth rinses and red food dye
* Dental prophylaxis within four weeks prior to Screening/Baseline 1 visit
* More than three sites that have periodontal pockets depths measuring 5mm or greater in depth
* Teeth having periodontal pocket depths measuring more than 3 mm in depth (healthy reference group)
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Use of Antibiotics, anti-inflammatory or anticoagulant therapy, phenytoin sodium or diphenylhydantoin, calcium channel blockers, cyclosporin A, immunostimulants/ immunomodulators during the study or within the one month prior to the Baseline 1 exam. Intermittent use of certain anti-inflammatory medication is acceptable at the discretion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Whole-mouth Mean Modified Gingival Index (Mean MGI) After 6 Weeks of Product Use | 6 weeks
  Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole-mouth Mean Plaque Index (Mean PI) After 6 Weeks of Product Use | 6 weeks
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).

SECONDARY OUTCOMES:
Whole-mouth Mean Plaque Index (Mean PI) After 4 Weeks of Product Use | 4 weeks
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).
Whole-mouth Mean Modified Gingival Index (Mean MGI) After 4 Weeks of Product Use | 4 weeks
  Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole-mouth Mean Expanded Bleeding Index (Mean BI) After 4 and 6 Weeks of Product Use | 4 and 6 Weeks
  Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 millimeter (mm) diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).
Percentage of Bleeding Sites, Based on the Expanded Gingival Bleeding Index After 4 and 6 Weeks of Product Use | 4 and 6 Weeks
  Percent bleeding sites will be calculated by taking the total number of sites with bleeding score greater than 0 divided by the total number of sites assessed for each participant. Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 millimeter (mm) diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Min K, Glowacki AJ, Bosma ML, McGuire JA, Tian S, McAdoo K, DelSasso A, Fourre T, Gambogi RJ, Milleman J, Milleman KR. Quantitative analysis of the effects of essential oil mouthrinses on clinical plaque microbiome: a parallel-group, randomized trial. BMC Oral Health. 2024 May 18;24(1):578. doi: 10.1186/s12903-024-04365-9. PMID 38762482
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSORC001793&attachmentIdentifier=7e32b18f-dbfa-4aed-8490-2a371807d184&fileName=CCSORC001793_Summary_CSR_Redacted.pdf&versionIdentifier=